CLINICAL TRIAL: NCT06182748
Title: Physical Activity and Fibrosing Interstitial Lung Disease
Acronym: AP-PID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230734
Record Dates: First submitted 2023-11-15; First posted 2023-12-27 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Fibrotic Interstitial Lungs Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training on eccentric ergocycle (experimental group) (Experimental): In eccentric cycling, pedals push against the user's feet in the opposite direction, user has to slow down pedals and quadriceps muscles lengthen during contraction.
  Interventions: Other: Training on eccentric ergocycle
- Training on concentric ergocycle (control group) (Active Comparator): In concentric cycling, quadriceps contract to push pedals.
  Interventions: Other: Training on concentric ergocycle

INTERVENTIONS:
Other: Training on eccentric ergocycle — Subjects will train on eccentric ergocycles. In eccentric cycling, pedals push against the user's feet in the opposite direction, user has to slow down pedals and quadriceps muscles lengthen during contraction.
  Other Names: Exercise training modality
  Arms: Training on eccentric ergocycle (experimental group)
Other: Training on concentric ergocycle — Subjects will train on regular concentric ergocycles. In concentric cycling, quadriceps contract to push pedals.
  Other Names: Exercise training modality
  Arms: Training on concentric ergocycle (control group)

SUMMARY:
Fibrotic interstitial lungs diseases (ILD) are a group of chronic and rare diseases characterized by an altered blood oxygenation in the lung, leading to dyspnea and physical limitation. Physical training is efficient to fight vicious circle of physical deconditioning observed in ILD. Eccentric cycling is an interesting modality of endurance training, allowing better exercise tolerance and adherence while developing cardiorespiratory function. Feasibility and efficacity of eccentric cycling were shown in chronic obstructive pulmonary disease but never in ILD. The primary aim of our work is to compare concentric and eccentric cycling training on physical capacities in ILD. Moreover, we will study the effects of training on the different steps of oxygen transport at exercise, from the lung to the muscles through the blood transport. Our second goal is then to characterize the physiological mechanisms underlying the benefits of exercising in ILD patients. Evaluations will be led during one year to study the long-term effects of training

DETAILED DESCRIPTION:
60 patients with fibrosing interstitial lung disease will be included in this study. Initial assessments at the beginning will be conducted for an overview of initials abilities and divided in 3 sessions. The first session (day 1) patients will be tested on maximal cardiopulmonary exercise testing with different devices to evaluate oxygen transport, and on different functional tests like 6minute walk test, sit to stand test, .. The second session (day 6) is composed by respiratory tests like spirometry, plethysmography and diffusing capacity of nitric oxyde and carbon monoxyde at rest and exercise. The last session, one week after the first (day 9), patients will performed a maximal cardiopulmonary treadmill testing, strength testing and physical activity questionnaire. Between day 1 and day 9, patients will be asked to wear an accelerometer to quantify daily physical activity and completed quality of life questionnaire. Then, patients will be randomised in control group (concentric cycling) and experimental group (eccentric cycling). They will be trained 3 times/week during 12 weeks at the same intensity, verified by gas exchange analysis (50 à 70% VO2reserve). The training is composed of aerobic training (eccentric or concentric cycling according to randomisation), muscle training and adapted sports. All assessments of the beginning will be also conducted after 12 weeks of training (3 months after inclusion) to study impact of training and between groups to compare the two cycling modalities in this population. To allow a follow-up after training, all assessments will be conducted 6 and 12 months after the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Fibrosing PID with fibrosis score > 10% of lung volume on chest CT scan
* Be able to attend physical reconditioning 3 times a week
* Be affiliated to a health insurance scheme
* Sign informed consent form

Exclusion Criteria:

* Any contraindication to physical activity (hereafter, after Dany-Michel Marcadeta, Bruno Pavy et al. Recommendations of the French Society of Cardiology for stress tests 2018)
* Be unable to perform exercise on an ergocycle or treadmill
* Be unable to perform a stress test, particularly for people on long-term oxygen therapy rest oxygen therapy at home
* IRS during an exacerbation
* Change in treatment < 3 months
* Sarcoidosis
* Connectivitis
* Pregnancy in progress
* Participation in a therapeutic intervention study
* Patient under guardianship
* Person subject to a legal protection measure
* Patient on state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2pic) during maximal cardiopulmonary exercise testing on ergocycle | VO2pic will be obtained at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  VO2pic is the gold standard indicator of cardiorespiratory function. In healthy people, disabled people and patients with ILD, there is a strong correlation between low VO2pic and high risk of mortality and comorbidities. It is often measured during incremental cardiopulmonary exercise testing with gas exchange measurements.Subjects have to cycle until exhaustion. VO2pic is the highest oxygen consumption recorded before test stop.

SECONDARY OUTCOMES:
During exercise testing : heart rate | All these evaluations will be obtained at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.
During exercise testing : ventilatory thresholds | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.
During exercise testing : power | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  power will be evaluated with handgrip test (number of repetition) Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population.
During exercise testing : speed | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  Distance walked (meters) Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population.
During exercise testing : distance covered on an inclined treadmill | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  distance covered on an inclined treadmill (meters) Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population.
During exercise testing : Cardiac output | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.
During exercise testing : muscular oxygenation | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  muscle oxygenation measured by near infrared spectroscopy (NIRS) (Oxygen quantity)
During exercise testing : blood gases | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  quantity of oxygen in arterial blood These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.
Functionnal fitness tests | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  number of chair lifts These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.
Physical activity : IPAQ (International Physical Activity Questionnaire) score | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.
Quality of life : SGRQ (ST. GEORGE'S RESPIRATORY QUESTIONNAIRE) score | at initial evaluation, after 3 months of training (M3), and 6 months and 12 months following the inclusion (M6 and M12, respectively)
  These evaluations show exhaustively different steps of oxygen transport, from breath to muscle extraction. Functionals tests show low level of physical fitness observed in ILD patients. Evaluation before and after training could show the impact of physical training on these parameters to improve quality of life and well being. In comparing different modalities of training, we would like to show what type of training is the most efficient for this population. As ILD patients have altered respiratory functions, evaluation before and after training could show improvement. General training can create neocapillarisation in muscle, we hypothesise that in the lung exercise training could conducted to a better diffusion in the lung, which is the core problem in fibrosing ILD.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise and Sports Medicine Department, Bobigny, Seine Saint Denis, France